CLINICAL TRIAL: NCT05923242
Title: Evaluation of Cardiovascular Health Outcomes Among Survivors 2 (ECHOS2) Pilot Intervention: Translating ECHOS Into an mHealth Platform
Brief Title: Translating ECHOS2 Into an mHealth Platform
Acronym: ECHOS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202305110
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Childhood Cancer; Cardiac Toxicity; Pediatric Cancer
Keywords: Anthracyclines; cardiotoxic therapy; chest radiation; mHealth; childhood cancer survivor; motivational interviewing
MeSH Terms: conditions — Neoplasms; Cardiotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerized Intervention Authoring Software (CIAS) (Experimental): Participants will be provided with a link to begin the study following consent, and the link will direct the participants to a baseline survey. At the end of the survey, participants will be automatically redirected to Computerized Intervention Authoring Software (CIAS). Participants will be encouraged to complete 2 sessions in CIAS, approximately 1 week apart. After completing the second session, CIAS will automatically redirect the participants to a post-test survey. Approximately 30 days after completing the second session, participants will be invited to complete a 30 day follow-up survey.
  Interventions: Behavioral: Computerized Intervention Authoring Software (CIAS)

INTERVENTIONS:
Behavioral: Computerized Intervention Authoring Software (CIAS) — CIAS is a web based intervention. The CIAS tool walks the participant through a Motivational Interviewing process whereby they think through the reasons for and against completing screening. CIAS makes use of an automated avatar (Emmi) who is programed to ask them questions and lead them through several topic areas related to screening. The CIAS pathways include options for participants to request a link of resources after they complete each session and for patients to request a list of the cancer treatments listed in their study records in order to confirm their understanding of their cancer history.

SUMMARY:
Childhood cancer survivors are at an increased risk of cardiac toxicity due to prior anti-cancer therapy. However, adherence to cardiac screening in this population remains low. This study aims to assess the feasibility of an mHealth motivational interviewing platform called Computerized Authoring Intervention Software (CIAS) in childhood cancer survivors. Participants will be recruited from the Childhood Cancer Survivorship Study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosed with cancer at age 17 or younger
* 2 or more years after completion of cancer therapy
* Receipt of cardiotoxic therapy (Any dose of anthracycline or 15 Gy chest radiation involving cardiac structures)
* No history of cardiomyopathy
* Have not received an echocardiogram in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in health belief model (HBM) construct scale of knowledge about echocardiograms and the effects of their treatment on health | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their knowledge of echocardiograms and the effects of their treatment on health on a 3 point scale consisting of possible answers of yes, no, and "don't know", with "don't know" being scored as incorrect. The scoring will be the summary of correct responses.
Change in self-determination theory (SDT) construct scale of competence, defined by confidence in getting an echocardiogram | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their confidence in getting an echocardiogram on a Likert scale with multiple choice between 0 to 10 with 0 indicating not at all sure and 10 indicating extremely sure. Scores will range from 0 and 10 with a higher value indicating higher confidence.
Change in self-determination theory (SDT) construct scale of autonomy, defined by the perceived choice of getting an echocardiogram | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their perceived choice of getting an echocardiogram on a 5-point Likert scale with 1 indicating disagree strongly and 5 indicating agree strongly. Scores will range from 3 to 15 with a higher score indicating higher perceived choice.
Change in self-determination theory (SDT) construct scale of relatedness, as defined by the effect of social norms/influence on the patient's decision of getting echocardiogram | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about the effects of social norms/influence on a 5-point Likert scale with 1 indicating disagree strongly and 5 indicating agree strongly. Scores will range from 6 to 30 with a higher score indicating more effect of social norms and influence on the patient's decision.
Change in movement toward screening | From post-test survey to 1 month follow-up (expected to be about 1 month and 1 week)
  Movement toward screening will consist of checking if patient made a plan to set an appointment with healthcare provider to discuss screening, made an appointment to discuss screening, had appointment to discuss screening, scheduled screening, or obtained screening, and if this plan changed between post-test survey and 1 month follow-up.

SECONDARY OUTCOMES:
Change in health belief model (HBM) construct scale of perceived risk of having heart problems | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their perceived risk of having heart problems on a 5 point scale, with 1 indicating no likelihood of heart problems, and 5 indicating extremely likely. Scores will range from 1 to 5 with a higher score indicating more perceived risk.
Change in health belief model (HBM) construct scale of perceived severity of having heart problems | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their perceived severity of heart problems on a 5 point scale, with 1 indicating not serious and 5 indicating extremely serious. Scores will range from 1 to 5 with a higher score indicating higher perceived severity.
Change in health belief model (HBM) construct scale of perceived barriers to getting echocardiogram | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their perceived barriers to getting an echocardiogram on a 5-point Likert scale with 1 indicating disagree strongly and 5 indicating agree strongly. Scores will range from 6 to 30 with a higher score indicating fewer perceived barriers.
Change in health belief model (HBM) construct scale of perceived benefits of getting echocardiogram | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their perceived benefits of getting an echocardiogram on a 5-point Likert scale with 1 indicating disagree strongly and 5 indicating agree strongly. Scores will range from 6 to 30 with a higher score indicating more perceived benefits.
Change in health belief model (HBM) construct scale of overall self-efficacy of getting echocardiogram | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their overall self-efficacy of getting an echocardiogram on a 5-point Likert scale with 1 indicating disagree strongly and 5 indicating agree strongly. Scores will range from 3 to 15 with a higher score indicating higher overall self-efficacy.
Change in health belief model (HBM) construct scale of worry about having heart problems | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their worry about having heart problems on a 5-point scale with 1 indicating not worried at all and 5 indicating extremely worried. Scores will range from 1 to 5 with a higher score indicating more worry.
Change in health belief model (HBM) construct scale intentions of getting echocardiogram | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their intentions of getting an echocardiogram on a 5-point Likert scale with 1 indicating disagree strongly and 5 indicating agree strongly. Scores will range from 3 to 15 with a higher score indicating a higher intention of getting an echocardiogram.
Change in self-determination theory (SDT) construct scale of intrinsic motivation, defined by the perceived importance of getting an echocardiogram | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their perceived importance of getting an echocardiogram on both a Likert scale with multiple choice between 0 to 10 with 0 indicating not at all important and 10 indicating extremely important, and a 5-point Likert scale with 1 indicating disagree strongly and 5 indicating agree strongly. Scores will range from 8 to 50 with a higher value indicating higher perceived importance.
Change in self-determination theory (SDT) construct scale of intrinsic motivation, defined by decision-making readiness | From baseline survey to post-test survey (expected to be about 1 week)
  Patients will be asked about their decision-making readiness in getting an echocardiogram on a Likert scale with multiple choice between 0 to 10 with 0 indicating not at all ready and 10 indicating extremely ready. Scores will range from 0 to 10 with a higher score indicating higher decision-making readiness.
Implementation process outcome of engagement with the app as measured by the time spent on the app | Through the second CIAS session (expected to be about 1 week)
  This will be defined as the total time spent on the app during session 1 and session 2.
Implementation process outcome of engagement with the app as measured by the number of modules started/completed | Through the second CIAS session (expected to be about 1 week)
  This will be defined as the total number of modules started and total number of modules completed on the app during session 1 and session 2.
Implementation process outcome of engagement with the app as measured by the number of sessions started/completed | Through the second CIAS session (expected to be about 1 week)
  This will be defined as the total number of sessions started and total number of sessions completed on the app during session 1 and session 2.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Waters, PhD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu